CLINICAL TRIAL: NCT06629623
Title: Current Status of Diagnosis, Treatment and Quality of Life for Patients with Idiopathic Pulmonary Fibrosis
Acronym: IPFLife
Status: Enrolling by invitation | Type: Observational
Sponsor: Chu Hongling (Other)
Collaborators: Boehringer Ingelheim (Industry); Beijing Chao Yang Hospital (Other); Zhejiang Chinese Medical University (Other Government); West China Hospital (Other); Peking University Shenzhen Hospital (Other)
Responsible Party: Sponsor-Investigator, Chu Hongling, Principal Investigator, Peking University Third Hospital
Organization: Peking University Third Hospital (Other)
Other Study IDs: M2024203
Record Dates: First submitted 2024-09-20; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic pulmonary fibrosis; rare disease; quality of life; mixed methods
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Rare Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with IPF
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The goal of this observational study is to explore current status of diagnosis, treatment and quality of life for patients with idiopathic pulmonary fibrosis. It aims to integrate qualitative and quantitative data to describe the distribution of perspective, experience, patient journey, treatment, expectation and quality of life for patients with idiopathic pulmonary fibrosis.

Participants will be invited to participate the interview, and answer quantitative survey questions about their quality of life.

DETAILED DESCRIPTION:
Idiopathic pulmonary fibrosis (IPF) is a rare, progressive, fibrotic interstitial lung disease of unknown aetiology primarily affecting middle-aged and elderly patients, more men than women. Median survival is 3∼5 years from the time of diagnosis. The prognosis is worse than for most common malignancies. However, patients' experiences, quality of life and needs during the disease course, have not been adequately investigated, which leads a lack of evidence to support the priority of treatment or drug development.

This study plans to conduct an mixed methods research to integrate qualitative and quantitative data to explore the perspective, experience, patient journey, treatment, expectation and quality of life for patients with idiopathic pulmonary fibrosis. For qualitative interview, there are 50 patients with idiopathic pulmonary fibrosis, and 15 physicians will be interviewed. For quantitative survey, there are 245 patients with idiopathic pulmonary fibrosis will be involved.

ELIGIBILITY:
Inclusion Criteria:

* IPF patients who are diagnosed according to international guidelines.
* Physicians who are clinical experts with extensive experience in the treatment of IPF.

Exclusion Criteria:

- The patient is unable to express his/her opinion clearly.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Under meeting the above inclusion and exclusion criteria, patients will be selected from Peking University Third Hospital, Beijing Chaoyang Hospital, Shenzhen Peking University-Hong Kong University of Science and Technology Medical Center, Zhejiang Chinese medical University, and West China Hospital of Sichuan University. Additionally, to ensure geographic representation of the patients, some participants will be recruited from a patient organization called "Take a Deep Breath for Love". A total of 295 IPF patients and 15 physicians are expected to represent six regions of the country, including Northeast, North China, Northwest, East China, Central South, and Southwest.
Sampling Method: Non-Probability Sample
Enrollment: 310 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Unmet patient needs | At beginning of study to explore by qualitative study, sequentially follow up at 6 month by quantitative survey
  Unmet patient needs primarily focus on the unmet clinical demands and expectations of IPF patients regarding their understanding and awareness of the disease, diagnosis, treatment methods, and patient management and care.
Patient journey | At beginning of study to explore by qualitative study, sequentially follow up at 6 month by quantitative survey.
  The patient journey primarily focuses on the entire process of IPF patients from the discovery of uncomfortable symptoms, diagnosis, and treatment to follow-up. By mapping the patient journey, we can identify the gaps between patients' expected experiences and their actual experiences at each stage, recognize and address common pain points, and gain insights into the value drivers behind patient decisions. This approach helps healthcare institutions to gain frontline perspectives on patient experiences in a timely manner, optimize disease diagnosis and treatment processes, develop scientifically sound treatment plans, and even assist in designing or enhancing mobile healthcare management solutions for patients.
Quality of life | At beginning of study to explore by qualitative study, sequentially follow up at 6 month by quantitative survey
  Quality of life primarily focuses on the impact of patients' physical and psychological health, as well as symptoms, and impact for their daily lives. Quality of life will be qualitatively deeply explore by interview, and quantitatively survey using EuroQol Five Dimensions Questionnair (EQ-5D) among patients with idiopathic pulmonary fibrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Hongling Chu, PhD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
This is a deeply exploration study about rare disease in China, which will integrate qualitative and quantitative data to answer the research question. This IPD data could not be shared. If some researchers plan to request IPD data, who could send email to the investigators. the investigators will review the request and send the available data.

REFERENCES:
- [Background] Kreuter M, Swigris J, Pittrow D, Geier S, Klotsche J, Prasse A, Wirtz H, Koschel D, Andreas S, Claussen M, Grohe C, Wilkens H, Hagmeyer L, Skowasch D, Meyer JF, Kirschner J, Glaser S, Herth FJF, Welte T, Neurohr C, Schwaiblmair M, Held M, Bahmer T, Frankenberger M, Behr J. Health related quality of life in patients with idiopathic pulmonary fibrosis in clinical practice: insights-IPF registry. Respir Res. 2017 Jul 14;18(1):139. doi: 10.1186/s12931-017-0621-y. PMID 28709421
- [Derived] Chu H, Ding Y, Zhou Y, Ji P, Yuan B, Zhan X, Lu X, Liu N, Zhang Y, Yan B, Fang X, Xu X, Huang Z, Li W, Shen N, Zhan S. Patient journey and Quality of Life for Patients with Idiopathic Pulmonary Fibrosis (IPFLife) in China: a sequential exploratory mixed methods research protocol. BMJ Open. 2025 Aug 12;15(8):e098770. doi: 10.1136/bmjopen-2025-098770. PMID 40803740